CLINICAL TRIAL: NCT02748291
Title: An Investigation Into the Role of Walking in Treating the Symptoms of Knee Osteoarthritis: The WalkOut Study
Acronym: WalkOut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Kimberley Edwards, Professor Sport Exercise & Nutrition Education, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G11122014 SoM ROD
Record Dates: First submitted 2016-04-15; First posted 2016-04-22 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis; Pain; Arthritis; Gonarthritis; Sedentary; Knee Osteoarthritis; Motor Activity; Physical Activity
Keywords: Sedentary; Knee osteoarthritis; Knee pain; Gonarthritis; Arthritis; Walking; Pedometer; Physical Activity; Activities of Daily Function; Department of Health Physical Activity Guidelines; Improve pain; Decrease pain; Improve function; Increase function; Activity Monitoring; Monitoring, Ambulatory/instrumentation
MeSH Terms: conditions — Osteoarthritis; Pain; Arthritis; Sedentary Behavior; Osteoarthritis, Knee; Motor Activity | interventions — Walking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walking (Experimental): Randomised participants will be instructed to walk 6,000 steps per day and throughout the day for 12 weeks. Step counts will be monitored by an issued pedometer. A 12 week paper diary will be provided for daily recording of step counts.
  Interventions: Other: Walking
- Control (Active Comparator): Department of Health (United Kingdom) Physical Activity Guidelines flyer (current standard of care).
  Interventions: Other: Department of Health Physical Activity Guidelines

INTERVENTIONS:
Other: Walking — The intervention group will be asked to walk a minimum 6,000 steps per day (7 days a week).
  Participants will be provided with a pedometer and daily diary to record step counts.
  Weekly scores will be collected via telephone contact.
  Followup questionnaires will be at 6, 12 and 24 months.
  Arms: Walking
Other: Department of Health Physical Activity Guidelines — 1. Adults should aim to be active daily. Over a week, activity should add up to at least 150 minutes (2½ hours) of moderate intensity activity in bouts of 10 minutes or more - one way to approach this is to do 30 minutes on at least 5 days a week.
  2. Alternatively, comparable benefits can be achieved through 75 minutes of vigorous intensity activity spread across the week or combinations of moderate and vigorous intensity activity.
  3. Adults should also undertake physical activity to improve muscle strength on at least two days a week.
  4. All adults should minimise the amount of time spent being sedentary (sitting) for extended periods.
  Arms: Control

SUMMARY:
There are over 8.75 million people in the United Kingdom with osteoarthritis in their knees. The effect of this condition can be debilitating. Symptoms are due to wear and tear of the knee joint. Some people can suffer with knee pain and stiffness. This study will look at whether walking improves the symptoms of knee osteoarthritis.

Investigators will recruit anyone with knee pain over the age of 45 years in Nottingham. Participants will undergo a full assessment by a qualified Doctor. After assessment, Participants meeting the eligibility criteria will be invited to join the study. Participants will be randomly allocated into 2 groups. One group will receive standard health and exercise advice. The other group will be allocated a walking activity. This group will undertake 6,000 walking steps each day. Participants will provide pedometers to monitor this walking activity.

The effect of walking will be compared using questionnaires. These will look at pain levels, quality of life and physical activity. The participants will complete these questionnaires before the study, at the 6 week midpoint and at the end of the 12 week intervention.

DETAILED DESCRIPTION:
BACKGROUND - Over 8.75 million people in the United Kingdom have painful osteoarthritis in one or both knees and a third of people of 45 years old have sought treatment. It has been well established that physical activity in mild - moderate osteoarthritis can provide improvement in symptoms and physical function. Current research is evaluating what modality of physical activity is best to achieve these improvements. A preliminary pedometer study in 2003 demonstrated symptomatic and functional improvement in knee osteoarthritis. A recent observational study has found that increased walking activity, with 6,000 steps per day being optimal, decreased the risk of functional limitation in knee osteoarthritis. Therefore, the purpose of this study is test evaluate the effectiveness of these recent recommendations against current UK physical activity guidelines.

AIMS - The study aims to investigate the role of walking in achieving a subjective improvement in symptomatic osteoarthritis of the knee/s. Furthermore, the study will investigate whether walking improves performance based tests which objectively assess physical function in participants with knee osteoarthritis. Null hypothesis to be tested: There is no difference in a 12 week intervention of walking 6,000 steps, per day, in improving pain and self reported physical function, compared to the current Department of Health physical activity guidelines.

EXPERIMENTAL PROTOCOL AND METHODS - Participants will be recruited through poster advertisement and non-incentivised involvement. Potential participants will be sent a Patient Information Leaflet for the study and a Consent Form. Following consent, the participant will be screened by telephone to ensure participants meet the inclusion criteria and also to exclude participants who would not be eligible on their medical history and activity status alone. Eligible participants from screening will be invited for a formal assessment. The assessment will confirm that information given in the screening remains accurate and a focussed physical examination of the knee. Participants eligible at the end of end of assessment will be randomly allocation into the control and intervention group, both lasting 12 weeks. Block randomisation will be used and this will be prepared by an independent person. Participants, irrespective of their allocation, will complete the following questionnaires: KOOS (KOOS: Knee Injury and Osteoarthritis Outcome Score), IPAQ (IPAQ: International Physical Activity Questionnaire), VAS for knee pain (VAS: Visual Analogue Scale), OKS (OKS: Oxford Knee Score), SF36 (SF36: Short Form Health Survey) and WOMAC (WOMAC: Western Ontario and McMaster Universities Arthritis Index). The intervention group will be allocated a walking activity of 6,000 per day. Participants will be provided with a pedometer and diary so walking activity can be recorded and monitored. Weekly scores will be collected via telephone contact with the participant. The control group will be provided with the standard physical activity advice that participants would receive from their GP (GP: General Practitioner) regarding physical activity levels. Both groups will complete a further IPAQ questionnaire at the mid point of the study at 6 weeks to monitor physical activity levels. At 12 weeks at the end of study, all participants will repeat the initial questionnaires, KOOS, IPAQ, VAS, OKS, SF36 and WOMAC and the performance based tests.

MEASUREABLE ENDPOINTS - Objective outcomes from performance based testing will be assessed, OARSI (OARSI: Osteoarthritis Research Society International) recommended physical function tests (6 minute walk test). Secondary outcomes: Pain, reported physical function in daily activities/sport/recreation, knee related quality of life measures from the above mentioned questionnaires and 4 other OARSI recommended functional tests (30sec chair stand test, 40m fast paced walk test, stair climb test and up and go test) in addition to age, sex, BMI (Body Mass Index), ethnicity and occupation.

N.B. 6,000 steps roughly equates to 2.5 miles/4.3 km. This distance is based on 71 steps to cover 100m (Investigator's 100m pace). At a steady pace, on flat terrain, 1 mile can be covered in 15minutes. The distance and timing to complete 6,000 steps will vary between participants depending on their stride length and pace.

ELIGIBILITY:
Inclusion Criteria:

Following current NICE (The National Institute for Health Care Excellence) guidelines (United Kingdom) for diagnosing knee osteoarthritis:

* Anyone over the age of 45 with painful knee/s
* No morning stiffness or stiffness that lasts less than 30 minutes

Exclusion Criteria:

* Exercise/activity > than current Department of Health physical activity guidelines
* Stiffness > 30mins in the morning
* Self-reported knee pathology (cruciate, meniscal, soft tissue, joint replacement)
* Cardiac disease - any:

  * Acute coronary syndrome < 12 months
  * Unexplained arrhythmia
  * Angioplasty/cardiac surgery
  * Congestive Cardiac Failure
  * Valvular disease
  * Cardiomyopathy
  * Myocarditis
  * Uncontrolled Hypertension
* Thrombolic events - any:

  * Cerebrovascular accident/transient ischaemic attack last 12 months
  * Deep vein thrombosis/pulmonary embolus last 6 months
* Asthma/Chronic Obstructive Pulmonary Disease Peak Expiratory Flow Rate < 300L/min/frequent exacerbations
* Anaemia Haemoglobin <90d/L
* Mental illness/learning disabilities/terminal illness
* Does not understand English

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Objective assessment of participant aerobic capacity and physical function measured in the 6 Minute Walk Test | 12 weeks

SECONDARY OUTCOMES:
Participant subjective opinion on their knee and associated symptoms measured by KOOS (Knee Injury and Osteoarthritis Score) | 12 weeks
Participant subjective opinion on their knee measured by WOMAC (Western Ontario and McMaster Universities Arthritis Index) Score | 12 weeks
Participant subjective opinion on their knee measured by OKS (Oxford Knee Score) | 12 weeks
Pain assessed VAS (Visual Analogue Scale) for knee pain | 12 weeks
Participant subjective opinion of their general and mental health assessed by SF36 (Short Form Health Survey) | 12 weeks
Objective assessment of participant physical function measured by OARSI (Osteoarthritis Research Society International) recommended functional tests for knee osteoarthritis - 30 second chair stand test | 12 weeks
Objective assessment of participant physical function measured by OARSI (Osteoarthritis Research Society International) recommended functional tests for knee osteoarthritis - 40 metre fast paced walk test | 12 weeks
Objective assessment of participant physical function measured by OARSI (Osteoarthritis Research Society International) recommended functional tests for knee osteoarthritis - stair climb test | 12 weeks
Objective assessment of participant physical function measured by OARSI (Osteoarthritis Research Society International) recommended functional tests for knee osteoarthritis - up and go test | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley L Edwards, MMedSci PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White DK, Tudor-Locke C, Zhang Y, Fielding R, LaValley M, Felson DT, Gross KD, Nevitt MC, Lewis CE, Torner J, Neogi T. Daily walking and the risk of incident functional limitation in knee osteoarthritis: an observational study. Arthritis Care Res (Hoboken). 2014 Sep;66(9):1328-36. doi: 10.1002/acr.22362. PMID 24923633
- [Background] Maddison R, Ni Mhurchu C, Jiang Y, Vander Hoorn S, Rodgers A, Lawes CM, Rush E. International Physical Activity Questionnaire (IPAQ) and New Zealand Physical Activity Questionnaire (NZPAQ): a doubly labelled water validation. Int J Behav Nutr Phys Act. 2007 Dec 3;4:62. doi: 10.1186/1479-5868-4-62. PMID 18053188
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Talbot LA, Gaines JM, Huynh TN, Metter EJ. A home-based pedometer-driven walking program to increase physical activity in older adults with osteoarthritis of the knee: a preliminary study. J Am Geriatr Soc. 2003 Mar;51(3):387-92. doi: 10.1046/j.1532-5415.2003.51113.x. PMID 12588583
- See also: Nice.org.uk, (2012). Walking and cycling: local measures to promote walking and cycling as forms of travel or recreation | Guidance and guidelines — http://www.nice.org.uk/guidance/ph41